CLINICAL TRIAL: NCT00171535
Title: A Study to Evaluate the Safety and Efficacy of Valsartan/Amlodipine Compared to Lisinopril/Hydrochlorothiazide Given Once Daily for 6 Weeks is Patients With Severe Hypertension
Brief Title: Efficacy and Safety of Valsartan/Amlodipine Combination in Patients With Severe Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAA489A2308
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2006-06

CONDITIONS: Hypertension
Keywords: hypertension; high blood pressure; valsartan; amlodipine
MeSH Terms: conditions — Hypertension | interventions — Amlodipine, Valsartan Drug Combination

INTERVENTIONS:
Drug: valsartan/amlodipine

SUMMARY:
This study will assess the effectiveness and safety of different combination antihypertensive treatments in patients with severe hypertension

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe hypertension

Exclusion Criteria:

* History of stroke, myocardial infarction, heart failure, chest pain, abnormal heart rhythm
* Liver, kidney, or pancreas disease
* Insulin dependent diabetes
* Allergy to certain medications used to treat high blood pressure

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2004-10; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Adverse events and serious adverse events at each study visit for 6 weeks

SECONDARY OUTCOMES:
Sitting and standing blood pressure measurements after 6 weeks
Laboratory test data after 6 weeks
Vital signs at each study visit for 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States